CLINICAL TRIAL: NCT02206295
Title: A Single-center, Open-label, Randomized, Two-period, Two-treatment, Crossover Study in Healthy Male Subjects to Demonstrate Bioequivalence of 1600 μg Selexipag Administered as Eight Tablets of 200 μg (Reference Drug) or as Single Tablet of 1600 μg (Test Drug)
Brief Title: Study in Healthy Male Subjects to Demonstrate Bioequivalence of 1600 μg Selexipag Administered as Eight Tablets of 200 μg or as Single Tablet of 1600 μg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-065-108
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Bioequivalence
Keywords: selexipag; ACT-333679
MeSH Terms: interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence AB (Experimental): Subjects will receive Treatment A in Period 1 followed by Treatment B in Period 2. There will be a washout period lasting at least 6 days between treatments.
  Treatment A: up-titration from Day 1-18 will performed in 200 μg steps every fourth day with multiples of 200 μg film-coated tablets starting with 400 μg selexipag b.i.d. The up-titration will be followed by treatment with 8 film-coated tablets, 200 μg each, b.i.d. from Day 19 to the morning dose of Day 23.
  Treatment B: up-titration from Day 1-18 will be performed in 200 μg steps every fourth day with multiples of 200 μg film-coated tablets starting with 400 μg selexipag b.i.d. The up-titration will be followed by treatment with one single film-coated tablet, 1600 μg, b.i.d. from Day 19 to the morning dose of Day 23.
  Interventions: Drug: selexipag
- Treatment Sequence BA (Experimental): Subjects will receive Treatment B in Period 1 followed by Treatment A in Period 2. There will be a washout period lasting at least 6 days between treatments.
  Treatment A: up-titration from Day 1-18 will performed in 200 μg steps every fourth day with multiples of 200 μg film-coated tablets starting with 400 μg selexipag b.i.d. The up-titration will be followed by treatment with 8 film-coated tablets, 200 μg each, b.i.d. from Day 19 to the morning dose of Day 23.
  Treatment B: up-titration from Day 1-18 will be performed in 200 μg steps every fourth day with multiples of 200 μg film-coated tablets starting with 400 μg selexipag b.i.d. The up-titration will be followed by treatment with one single film-coated tablet, 1600 μg, b.i.d. from Day 19 to the morning dose of Day 23.
  Interventions: Drug: selexipag

INTERVENTIONS:
Drug: selexipag

SUMMARY:
The primary aim of this study is to demonstrate bioequivalence in the rate and extent of absorption between 1600 μg selexipag test drug (administered orally as film-coated tablets of 1600 μg, twice a day (b.i.d.) and 1600 μg selexipag reference drug (administered orally as 8 film-coated tablets of 200 μg b.i.d.) at steady-state in healthy male subjects following a multiple-dose up-titration scheme.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Healthy male subjects aged between 18 and 55 years (inclusive) at Screening.
* No clinically significant findings on the physical examination at Screening.
* Body mass index of 18.0 to 30.0 kg/m^2 (inclusive) at Screening.
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 beats per minute (all inclusive), measured at Screening.
* 12-lead electrocardiogram without clinically relevant abnormalities, measured at Screening.
* Hematology, clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent at Screening.
* Negative results from urine drug screen and alcohol breath test at Screening.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known allergic reactions or hypersensitivity to selexipag or any excipient of the drug formulation used in this study.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of selexipag.
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
* Treatment with selexipag or another investigational drug within 1 month prior to Screening or 5 half-lives, whichever is longer.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening.
* Excessive caffeine consumption at Screening.
* Smoking within 3 months prior to Screening and inability to refrain from smoking during the course of the study.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter medications within 2 weeks prior to first study drug administration.
* Loss of 500 mL or more of blood within 3 months prior to Screening.
* Positive results from the hepatitis serology (hepatitis B antigen and hepatitis C antibodies), except for vaccinated subjects or subjects with past but resolved hepatitis, at Screening.
* Positive results from the human immunodeficiency virus serology at Screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at Screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUCt) for selexipag | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. Selexipag will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. AUCt will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification during one dosing interval.
Maximum plasma concentration at steady state (Cmax,ss) for selexipag | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. Selexipag will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. The measured individual plasma concentrations of selexipag will be used to directly obtain Cmax,ss.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUCt) for ACT-333679 | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. ACT-333679 will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. AUCt will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification during one dosing interval.
Maximum plasma concentration at steady state (Cmax,ss) for ACT-333679 | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. ACT-333679 will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. The measured individual plasma concentrations of ACT-333679 will be used to directly obtain Cmax,ss.
Time to reach maximum plasma concentration at steady state (tmax,ss) for selexipag | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. Selexipag will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. The measured individual plasma concentrations of selexipag will be used to directly obtain tmax,ss.
Trough plasma concentration at the end of one dose interval (Ctrough) for selexipag | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. Selexipag will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. The measured individual plasma concentrations of selexipag will be used to directly obtain Ctrough.
Trough plasma concentration at the end of one dose interval (Ctrough) for ACT-333679 | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. ACT-333679 will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. The measured individual plasma concentrations of ACT-333679 will be used to directly obtain Ctrough.
Trough plasma concentration at steady state (Ctrough,ss) for selexipag | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. Selexipag will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. The measured individual plasma concentrations of selexipag will be used to directly obtain Ctrough,ss.
Trough plasma concentration (Ctrough,ss) for ACT-333679 | 23 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in an arm vein after 4.5 days' treatment with 1600 μg selexipag b.i.d. during Treatments A and B. ACT-333679 will be quantified in plasma samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) assay. The measured individual plasma concentrations of ACT-333679 will be used to directly obtain Ctrough,ss.
Change in systolic blood pressure from baseline up to end of study | up to 28 days
  Blood pressure and pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand).
Change in diastolic blood pressure from baseline up to end of study | up to 28 days
  Blood pressure and pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand).
Change in pulse rate from baseline up to end of study | up to 28 days
  Blood pressure and pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand).
Change in body weight from baseline up to end of study | up to 28 days
  Blood pressure and pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand).
Change in heart rate from baseline up to end of study | up to 28 days
  Heart rate will be measured using standard 12-lead electrocardiography recorded at rest with the subject in the supine position for a 5 minute period.
Change in PQ/PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) from baseline up to end of study | up to 28 days
  PQ/PR interval will be measured using standard 12-lead electrocardiography recorded at rest with the subject in the supine position for a 5 minute period.
Change in QRS interval (time interval from the beginning of the Q wave to the end of the S wave) from baseline up to end of study | up to 28 days
  QRS interval will be measured using standard 12-lead electrocardiography recorded at rest with the subject in the supine position for a 5 minute period.
Change in QT interval (time interval from beginning of the Q wave until end of the T wave) from baseline up to end of study | up to 28 days
  QT interval will be measured using standard 12-lead electrocardiography recorded at rest with the subject in the supine position for a 5 minute period.
Change in QTcB interval (time interval from beginning of the Q wave until end of the T wave, according to Bazett's correction) from baseline up to end of study | up to 28 days
  QT interval will be measured using standard 12-lead electrocardiography recorded at rest with the subject in the supine position for a 5 minute period. QTcB will be calculated according to the following formula (QTcB = QT/RR^0.5 where RR is 60/heart rate).
Change in QTcF interval (time interval from beginning of the Q wave until end of the T wave, according to Fridericia's correction) from baseline up to end of study | up to 28 days
  QT interval will be measured using standard 12-lead electrocardiography recorded at rest with the subject in the supine position for a 5 minute period. QTcF will be calculated according to the following formula (QTcF = QT/RR^0.33 where RR is 60/heart rate).
Number of treatment-emergent electrocardiogram abnormalities from baseline up to end of study | up to 28 days
  Electrocardiogram abnormalities will be measured using standard 12-lead electrocardiography recorded at rest with the subject in the supine position for a 5 minute period.
Number of participants with adverse events leading to discontinuation of study treatment | up to 28 days
  Adverse events will be considered as any adverse change from the subject's baseline condition that occurred during the course of the study. The subjects will be required to report any adverse events spontaneously. In addition, each subject will be assessed by the investigator at any measurement timepoint as well as at the end of observation and whenever necessary as deemed by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Baldoni, PhD, PharmD, Study Director — Actelion